CLINICAL TRIAL: NCT06991361
Title: A Phase I Trial of Ex Vivo-Expanded (EVE) Regulatory T Cells in Combination With Low-Dose Interleukin-2 for Steroid-Refractory Chronic Graft-versus-Host-Disease
Brief Title: Ex Vivo-Expanded Regulatory T Cells Plus Low-Dose Interleukin-2 for Steroid-Refractory Chronic GVHD
Acronym: EVENT
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Leslie Kean (Other)
Responsible Party: Sponsor-Investigator, Leslie Kean, Director, Stem Cell Transplant Program, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00025318
Record Dates: First submitted 2025-05-20; First posted 2025-05-27 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Graft Versus Host Disease (cGvHD)
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level A (Experimental): EVE Treg Cell dose level A
  Interventions: Biological: EVE-Treg
- Dose Level B (Experimental): EVE Treg Cell dose level B
  Interventions: Biological: EVE-Treg
- Dose Level C (Experimental): EVE Treg Cell dose level C.
  Interventions: Biological: EVE-Treg

INTERVENTIONS:
Biological: EVE-Treg — Ex Vivo-Expanded (EVE) Regulatory T cells.

SUMMARY:
Hematopoietic Stem Cell Transplant (HCT) has been used to treat children and adults who have leukemia, lymphoma and other cancers of blood and immune cells since the 1970s. For many of these forms of cancer, HCT works well. However, HCT can cause serious, sometimes life-threatening complications.

One of the most serious and common complications of HCT is graft-versus-host disease (GVHD). GVHD can appear early after the transplant, usually about 3 to 4 weeks after the transplant is given. This is called acute GVHD (aGVHD), because it usually happens over a couple of days. If successfully treated, acute GVHD quickly goes away. Sometimes GVHD happens months after the transplant. Then it is called chronic GVHD (cGVHD), because it happens gradually and goes away slowly.

The investigators are doing this study to see if one dose of Ex vivo-Expanded Regulatory T cells (EVE-Treg) can be used together with the daily Interleukin 2 (IL-2) to treat cGVHD, that has not responded to steroid treatment or low-dose IL-2.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of 7-8/8 HLA-matched allogeneic hematopoietic stem cell transplantation or recipient of haploidentical allogenic hematopoietic stem cell transplantation.
* Age 2 and up.
* Must have steroid-refractory chronic GVHD that is still active despite at least 4 weeks of treatment with low-dose subcutaneous (SC) IL-2.
* Stable dose of glucocorticoids for 2 weeks prior to enrollment
* no addition or subtraction of other immunosuppressive medications for 4 weeks prior to enrollment.
* Must have adequate organ and marrow function.
* Ability to understand and willingness to sign a written informed consent form.
* Donor who is willing and cleared to donate starting material for manufacture of EVE-Treg.

Exclusion Criteria:

* Recipient of umbilical cord blood stem cell graft.
* Ongoing prednisone requirement greater than 1 mg/kg/day (or equivalent).
* Karnofsky/Lansky performance score less than 40%.
* Concurrent use of methotrexate, azathioprine, or a calcineurin-inhibitor plus sirolimus.
* Other investigational agents within 4 weeks prior to enrollment.
* Participants with post-transplant exposure to donor lymphocyte infusion, or T-cell or IL-2 targeted medications within 100 days prior to enrollment.
* Participants with new immunosupprssive medication, extra-corporeal photopheresis or rituximab therapy initiated int he 4 weeks prior to enrollment.
* Participants with active malignant relapse or recrudescence of their prior hematologic disorder.
* Uncontrolled intercurrent illness unrelated to cGVHD.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant patients are excluded.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety of EVE-Treg | 5 weeks
  Safety of EVE-Treg, in combination with physician-prescribed daily low-dose IL-2, for the treatment of chronic GVHD refractory to steroids and low-dose IL-2. Safety will be based on adverse events at each Dose Level of EVE-Treg

IPD SHARING:
Plan to Share IPD: Undecided